CLINICAL TRIAL: NCT07231705
Title: Growth and Enteral Tolerance of Plant-Based Enteral Formulas: A Prospective Study
Brief Title: Growth and Tolerance of Plant-based Enteral Formulas in Children Ages 12-17 Months.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kate Farms Inc (Industry)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nationwide2025
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Formula Dependent Children 1 to 2 Years of Age

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formula (Experimental): The study intervention will be 2 pea protein-based formulas Kate Farms Pediatric Standard formula 1.2 (KF-PS) and Kate Farms Standard Pediatric Peptide Formula 1.0 (KF-PP).
  Interventions: Dietary Supplement: Kate Farms Standard 1.2 or Peptide 1.0

INTERVENTIONS:
Dietary Supplement: Kate Farms Standard 1.2 or Peptide 1.0 — Kate Farms Standard 1.2 or Peptide 1.0 formulas will be provided by mouth or via tubefeeding. Study children will be fed the formula for a period of up through 24 weeks.

SUMMARY:
The purpose of this prospective study is to evaluate the growth and enteral tolerance of two pea protein-based formulas from Kate Farms in children aged 12 to 17 months who are expected to meet most of their nutritional needs through formula. It is hypothesized that the Pediatric Standard 1.2 and Pediatric Peptide 1.0 formulas will support healthy growth in children between 1 and 2 years of age. The study will assess the impact of these formulas on growth, tolerance, body composition, micronutrient levels, and gut microbiome health in tube-fed children. Formula will be provided for 24 weeks.

DETAILED DESCRIPTION:
This is a prospective cohort study. Forty children ages 12-17 months who rely on formula for at least 80% of their nutritional needs (by mouth of tube feeding) are expected to continue this dependence for the next 6 months will be recruited. Children will be recruited from the Feeding Program, GI clinic and Complex Care clinic at Nationwide Children's Hospital in Columbus, Ohio. The study will be introduced to the patient by the provider during a routine clinic visit. Parent consent will be obtained from one of the research investigators during the clinic visit.

The objectives are to study the effect of these formulas on the functions of the body (AND NOT to evaluate its role in any disease state) in the form of growth and nutrition status.

- To sustain/improve to a weight-for-length z-score of between -1 and 0 up through 24 weeks, in children who are predominantly receiving nutrition via formula (either orally or via tube feeding)

Secondary study objectives:

* To sustain other anthropometric measurements
* To assess tolerance
* To assess changes in body composition and gut microbiome
* To assess changes in key micronutrients.

To sustain the following z scores up through 24 weeks relative to baseline:

* Weight-for-age
* Length-for-age
* Head circumference-for-age
* Mid upper arm circumference (MUAC)-for-age
* Weight velocity
* Length velocity o When ex-preterm infants are recruited, all of these measures will be corrected for gestational age.

Tolerance: Composite measure of tolerance using 3-day diaries:

* Percentage of feedings that result in spit up/vomiting
* Average number of stools/day
* Average stool consistency score using the Brussels Infant and Toddler stool scale
* Gastrointestinal and Gastroesophageal Reflux (GIGER) Scale for Infant and Toddlers

Body composition: Bioelectrical impedance analysis Gut microbiome: Stool microbiome analysis Micronutrient analysis: Iron and zinc nutriture

ELIGIBILITY:
Inclusion Criteria:

* Children, male or female, aged 12 through 17 months (for premature infants, we will use corrected age)
* Children with a weight-for-length z score between ≥ -1.5 at enrolment
* Children obtaining via formula feeding ≥ 80% of their total energy intake at enrolment and expected to continue to require such formula intake for the next 24 weeks
* Children from families who are willing and able to comply with the requirements of the protocol
* Written informed consent from the parent or legal guardian
* Parent/caregiver or legal guardian must be able to read, write, and understand English

Exclusion Criteria:

* Children with known or suspected complex gastrointestinal anomalies or dysfunction, hepatic or renal dysfunction, or inherited metabolic disorders, suspected or diagnosed conditions associated with malabsorption (e.g. cystic fibrosis) (Note: For hepatic dysfunction, a conjugated bilirubin >2.0 mg/dL and for renal dysfunction child should not meet any of the Pediatric Risk, Injury, Failure, Loss, End Stage Renal Disease (pRIFLE) criteria for renal disease (estimated creatinine clearance decreased by 25% by the Schwartz formula or urine output <0.5 mL/kg per hour over the previous 8 or more hours) or has chronic medical renal disease. We will not obtain labs to exclude children. If children are noted to have liver disease or renal disease in their chart, we will look at their labs to ensure that they do not meet exclusion criteria).
* Children with tracheostomy and/or inspired oxygen via nasal cannula or children receiving diuretics.
* Children with known or suspected genetic and/or metabolic inborn errors of metabolism conditions known to interfere with growth or body dysmorphology that can interfere with obtaining standard anthropometric measurements (weight, length, head circumference, and arm circumference)
* At study entry, children expected to consume on average more than 20% of their energy intake from non-formula sources of nutrition: solids, expressed breast milk and /or parenteral nutrition.
* Child requiring or expected to have an energy requirement < 80 kcal/kg per day - Breastfeeding child (who is feeding at the breast > 2 times per day)
* Child likely to undergo major surgery during the duration of the study
* Child with a nasogastric tube that is unlikely to get a gastrostomy tube during the duration of the study
* Principal Investigator's uncertainty about the willingness or ability of the parent/caregiver to comply with the protocol requirements
* Children whose parent is younger than the legal age of consent
* Children with known allergy to pea protein or soy or peanuts.
* Children with a parent or a sibling with a known allergy to pea protein or soy or peanuts.

Ages: 12 Months to 17 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Weight-for-length z-score | 24 weeks
  To sustain/improve to a weight-for-length z-score of between -1 and 0 up through 24 weeks, in children who are predominantly receiving nutrition via formula (either orally or via tube feeding)

SECONDARY OUTCOMES:
Weight-for-age | 24 weeks
  Z-scores for weight-for-age of between -1 and 0 up through 24 weeks relative to baseline.
Length-for-age | 24 weeks
  Z scores for length-for-age of between -1 and 0 up through 24 weeks relative to baseline.
Head circumference-for-age | 24 weeks
  Z-scores for head circumference-for-age of between -1 and 0 up through 24 weeks relative to baseline.
Mid upper arm circumference (MUAC)-for-age | 24 weeks
  Z-scores for mid upper arm circumference (MUAC)-for-age of between -1 and 0 up through 24 weeks relative to baseline.
Weight velocity | 24 weeks
  Average weight velocity in grams (g)
Length velocity | 24 weeks
  Average length velocity in centimeters (cm)
Tolerance - Spit up/vomiting | 24 weeks
  Percentage of feedings that results in spit up/vomiting based on 3-day food diaries
Tolerance - Stool | 24 weeks
  Average number of stools per day
Tolerance - Stool consistency | 24 weeks
  Average stool consistency using the Brussels Infant and Toddler Stool Scale
Gastrointestinal (GI) and gastroesophageal (GER) reflux symptoms | 24 weeks
  GI and GER symptoms using the Gastrointestinal and Gastroesophageal Reflux (GIGER) Scale for Infants and Toddler
Body Composition | 24 weeks
  Body composition parameters using a bioelectrical impedance analysis
Gut Microbiome | 24 weeks
  Stool microbiome analysis
Micronutrient analysis | 24 weeks
  Iron and zinc nutriture

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Goday, MD, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No